CLINICAL TRIAL: NCT02978729
Title: A Randomized Study of Telephone Versus Videoconference Communication for Remote Genetic Disclosure in the APOE4 Trial
Brief Title: Telephone Versus Videoconference Communication for Remote Genetic Disclosure in the APOE4 Trial
Acronym: CONNECT4APOE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 824225
Record Dates: First submitted 2016-11-07; First posted 2016-12-01 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Alzheimer Disease; Genetic Predisposition to Disease
Keywords: Telemedicine; Counseling, Genetic
MeSH Terms: conditions — Alzheimer Disease; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone (Active Comparator): Telephone telegenetics counseling: A trained Penn genetic counselor will conduct genotype disclosure visits with the participant via telephone. The participant will be in a private room at the study site. Telephone sessions will utilize a private phone line. The genetic counselor will use standardized disclosure checklist and visual aids for the disclosure session.
  Interventions: Other: Telephone remote genetic counseling
- Videoconference (Experimental): Two-way videoconferencing telegenetics counseling: A trained Penn genetic counselor will conduct genotype disclosure visits with the participant via two-way videoconferencing. The participant will be in a private room at the study site. Videoconferencing sessions will utilize tablets or laptops with web cameras and secure/confidential software for teleconferencing. The genetic counselor will use standardized disclosure checklist and visual aids for the disclosure session.
  Interventions: Other: Two-way videoconference remote genetic counseling

INTERVENTIONS:
Other: Two-way videoconference remote genetic counseling
  Arms: Videoconference
Other: Telephone remote genetic counseling
  Arms: Telephone

SUMMARY:
The purpose of this study is to compare two methods for remote genetic counseling (telephone and two-way videoconferencing) for patients who are receiving disclosure of their APOE (apolipoprotein E) genotype. The target population will consist of males and females in the age range of 60-75 years who, as potential participants in a study (Generation Study), will need to receive genetic counseling and disclosure of APOE genotype. Subjects must be willing to receive genetic counseling and disclosure remotely. Subjects must be willing to be randomized to either telephone arm or videoconference arm.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible to participate in the Generation Study
2. Ability to provide consent
3. Ability to communicate and hear in English

Exclusion Criteria:

-

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2016-08; Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Satisfaction with genetic counseling services as measured by the Satisfaction with Genetic Services Scale | 2-7 days
Satisfaction with genetic counseling services as measured by the Satisfaction with Remote Counseling Scale | 2-7 days

SECONDARY OUTCOMES:
Knowledge of Genetic Disease as measured by the Cancer Genetics Knowledge Scale | 2-7 days, 6 weeks, 6 months, 12 months
Disease-specific distress as measured by the Impact of Events Scale | 2-7 days, 6 weeks, 6 months, 12 months
Perceived risk of Alzheimers Disease as measured by questionnaire items measuring perceived risk in quantitative, qualitative, and relative terms | 2-7 days, 6 weeks, 6 months, 12 months
Responses to Genetic Testing as measured by the Impact of Genetic Testing for Alzheimer's disease (IGT-AD) scale | 2-7 days, 6 weeks, 6 months, 12 months
Depression as measured by the GDS Short Form | 2-7 days, 6 weeks, 6 months, 12 months
Anxiety as measured by the Mini State Trait Anxiety Inventory (mSTAI): | 2-7 days, 6 weeks, 6 months, 12 months
Knowledge of Genetic Disease as measured by the ClinSeq Knowledge Scale | 2-7 days, 6 weeks, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Angela R Bradbury, MD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No